CLINICAL TRIAL: NCT03499210
Title: A Multi-site, Interventional, Non-comparative, Single-arm Trial to Evaluate the Safety of the ReWalk ReStore Device in Subjects With Mobility Impairments Due to Ischemic or Hemorrhagic Stroke
Brief Title: Safety Evaluation of the ReWalk ReStore Device in Subjects With Mobility Impairments Due to Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ReWalk Robotics, Inc. (Industry)
Collaborators: Shirley Ryan AbilityLab (Other); Kessler Foundation (Other); TIRR Memorial Hermann (Other); Spaulding Rehabilitation Hospital (Other); Moss Rehabilitation Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLN0011
Record Dates: First submitted 2018-03-27; First posted 2018-04-17 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Stroke; Stroke, Acute; Stroke Hemorrhagic; Hemiparesis; Hemiplegia; Cerebrovascular Accident
Keywords: Stroke; Exoskeleton; Hemiparesis; Hemiplegia
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Investigational group (Experimental): All subjects will participate in study procedures involving use of the ReWalk ReStore device.
  Interventions: Device: ReWalk ReStore device

INTERVENTIONS:
Device: ReWalk ReStore device — The ReWalk ReStore device is intended to be used to perform ambulatory functions in rehabilitation institutions under the supervision of a trained therapist for people with hemiplegia/hemiparesis due to stroke.

SUMMARY:
A multi-site, interventional, non-comparative, single-arm trial to evaluate the safety of the ReWalk ReStore device in subjects with hemiplegia/hemiparesis due to ischemic or hemorrhagic stroke.

ELIGIBILITY:
Inclusion Criteria:

* History of one-sided ischemic or hemorrhagic stroke (>2 weeks post stroke)
* Presentation of hemiparesis/hemiplegia resulting from stroke
* At least 18 years of age
* Height of 4'8" - 6'7"
* Weight of less than 264 lbs
* Medical clearance by a clinician treating the subject
* Able to ambulate at least 5 feet without an ankle foot orthosis (AFO), with no more than minimal contact assistance from a PT
* Able to follow a 3-step command
* Able to fit suit components (waistbelt, calf wrap)
* No greater than 5 degrees of plantar flexion contracture during passive ankle ROM
* Modified Ashworth Scale for spasticity at 3 or less for ankle dorsi-flexors and plantar-flexors

Exclusion Criteria:

* Severe aphasia limiting ability to express needs or discomfort verbally or non-verbally
* Serious co-morbidities that, in the opinion of the investigator, may interfere with ability to participate
* History of significant Peripheral Artery Disease
* Colostomy bag
* Current pregnancy
* Uncontrolled or untreated hypertension
* Currently participating in any other ongoing clinical trial
* Presence of open wounds or broken skin at device locations requiring medical management
* Known urethane allergies
* Current medical diagnosis of DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related adverse events [Safety] | duration of study participation for each subject, estimated 4 weeks
  Safety will be evaluated on the basis of the number of device-related adverse events reported for subjects during their participation in the study.

SECONDARY OUTCOMES:
Incidence of device malfunctions during study procedures [Device Reliability] | duration of study completion for each site, estimated 4 months
  Device reliability will be evaluated on the basis of the number of device malfunctions reported by research study staff for the duration of study procedures at each study site.
Incidence of injury to physical therapist caused by device [PT safety] | duration of study completion for each site, estimated 4 months
  PT safety will be evaluated on the basis of the number of device-related injuries reported by study physical therapists for the duration of study procedures at each study site.

OTHER OUTCOMES:
Gait speed measured with 10 Meter Walk Test | duration of study participation for each subject, estimated 4 weeks
  Subjects will perform a 10 Meter Walk Test to evaluate walking speed with and without the ReStore device.
Gait analysis using a gait mat | duration of study participation for each subject, estimated 4 weeks
  Subjects will walk across a gait mat device (such as GAITRite) which records step timing and step placement in order to evaluate their walking with and without the ReStore device.
Walking distance measured with 2 Minute Walk Test | duration of study participation for each subject, estimated 4 weeks
  Subjects will perform a 2 Minute Walk Test (2MWT) to evaluate the 2 minute walking distance with the ReStore device in Slack, Assist, and Brace modes
Modified QUEST questionnaire [subject satisfaction] | duration of study participation for each subject, estimated 4 weeks
  Subjects will complete a modified QUEST questionnaire (Quebec User Evaluation of Assistive Technology) to indicate their level of satisfaction with the ReStore device (on a scale from 1 to 5) in 8 different categories.
Physical Therapist satisfaction questionnaire [PT satisfaction] | duration of study completion for each site, estimated 4 months
  Physical Therapists involved in the study will complete a PT satisfaction questionnaire at the end of the study to indicate their level of satisfaction (on a scale from 1 to 5) with the ReStore device in 9 different categories.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Spaulding Rehabilitation Institute, Boston, Massachusetts
  - Kessler Foundation, West Orange, New Jersey
  - Moss Rehab, Elkins Park, Pennsylvania
  - TIRR Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Awad LN, Esquenazi A, Francisco GE, Nolan KJ, Jayaraman A. The ReWalk ReStore soft robotic exosuit: a multi-site clinical trial of the safety, reliability, and feasibility of exosuit-augmented post-stroke gait rehabilitation. J Neuroeng Rehabil. 2020 Jun 18;17(1):80. doi: 10.1186/s12984-020-00702-5. PMID 32552775